CLINICAL TRIAL: NCT00860184
Title: Assessment of MRI-based Prediction of Stroke and Other Cerebrovascular Symptoms Arising From Carotid Atherosclerotic Disease in Asymptomatic Individuals
Brief Title: SmartRisk Stroke Prediction by MRI of Carotid Disease
Acronym: SmartRisk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: VPDiagnostics (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: William Kerwin / Vice President of Research and Development, VPDiagnostics, Inc.
Other Study IDs: VPD2008A; 5R44HL070576-05 (NIH)
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Atherosclerotic Disease, Carotid
Keywords: carotid artery; atherosclerosis; stroke; transient ischemic attack; MRI; software; risk
MeSH Terms: conditions — Carotid Artery Diseases; Atherosclerosis; Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 50-79% stenosis: Subjects with 50-79% stenosis of the carotid artery Absence of prior ischemic neurological symptoms Age 18 or older

SUMMARY:
Atherosclerotic plaque at the carotid artery bifurcation is a major source of stroke. The purpose of this investigation is to determine the ability of the SmartRisk software module to predict stroke or stroke-related events due to carotid plaque within a high-risk population. The SmartRisk software module operates on magnetic resonance images (MRI) of the carotid artery wall.

DETAILED DESCRIPTION:
Carotid artery disease (atherosclerosis) is a major cause of stroke that can be treated with carotid endarterectomy surgery (CEA) or stenting. Subjects with moderate, asymptomatic stenosis (50-79% narrowing) typically do not undergo intervention because the procedural risks outweigh the benefits. However, some of these individuals will have vulnerable plaque that places them at high risk of stroke, but current diagnostic techniques for vulnerable plaque are lacking. Recently, VPDiagnostics developed a new module - SmartRisk - that stratifies risk of stroke for stenotic (50-79% blockage) atherosclerotic plaque. The SmartRisk module uses MRI data to compute a risk assessment from a specific atherosclerotic plaque. A continuous risk value is generated and patients with risk values above a prespecified threshold are at elevated risk for cerebrovascular events arising from carotid artery disease. The purpose of this trial is to determine whether the SmartRisk module is effective at stratifying risk of a carotid-related cerebrovascular event in subjects with asymptomatic 50-79% carotid stenosis.

ELIGIBILITY:
Inclusion Criteria:

* 50-79% stenosis of the carotid artery
* age 18 or older
* no ischemic neurovascular symptoms within preceding 6 months

Exclusion Criteria:

* contraindication to MRI (e.g. weight > 130 kg, pregnancy)
* prior or planned carotid endarterectomy or stenting
* history of atrial fibrillation
* prior neck irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient referred for ultrasound assessment of carotid artery disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
stroke or other cerebrovascular symptom (e.g. TIA) | 18 month mean follow-up at 6 month intervals

SECONDARY OUTCOMES:
any cardiovascular event (e.g. MI) | 18 month mean follow-up at 6 month intervals

CONTACTS AND LOCATIONS:
Overall Officials: William S Kerwin, PhD, Principal Investigator — VPDiagnostics
Locations (15):
- United States (15):
  - Carl T. Hayden Medical Research Foundation, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Gotham Cardiovascular Research PC, New York, New York
  - New York University School of Medicine, New York, New York
  - Baylor College of Medicine, Houston, Texas
  - Western Institute for Biomedical Research, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- See also: VPDiagnostics website — http://www.vpdiagnostics.com